CLINICAL TRIAL: NCT02776813
Title: Phase 1 Study of ACTR087, Autologous T Lymphocytes Expressing Antibody Coupled T-cell Receptors (CD16V-41BB-CD3ζ), in Combination With Rituximab, in Subjects With Relapsed or Refractory CD20-Positive B-Cell Lymphoma
Brief Title: Study of ACTR087 in Subjects With Relapsed or Refractory B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UT-201501; ATTCK-20-2 (Other: Unum Therapeutics)
Record Dates: First submitted 2016-05-04; First posted 2016-05-18 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: CD20+; B-cell; ACTR087; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACTR087, in combination with rituximab (Experimental)
  Interventions: Biological: ACTR087; Biological: rituximab

INTERVENTIONS:
Biological: ACTR087
Biological: rituximab

SUMMARY:
This is a phase 1, multi-center, single-arm, open-label study evaluating the safety and efficacy of an autologous T-cell product expressing ACTR in combination with rituximab in subjects with refractory or relapsed CD20+ B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures
* Histologically-confirmed relapsed or refractory CD20+ B-cell lymphoma of one of the following types, with documented disease progression or recurrence following the immediate prior therapy:

  * DLBCL, regardless of cell of origin or underlying molecular genetics
  * MCL
  * PMBCL
  * Gr3b-FL
  * TH-FL
* Biopsy-confirmed CD20+ expression of the underlying malignancy by immunohistochemical staining or flow cytometry between the most recent dose of an anti-CD20 monoclonal antibody (mAb) and study enrollment
* At least 1 measurable lesion on imaging. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
* Must have received adequate prior therapy for the underlying CD20+ B-cell lymphoma, defined as an anti-CD20 mAb in combination with an anthracycline-containing chemotherapy regimen (i.e. chemo-immunotherapy) and at least one of the following:

  * biopsy-proven refractory disease after frontline chemo-immunotherapy
  * relapse within 1 year from frontline chemo-immunotherapy and ineligible for autologous hematopoietic stem cell transplant (auto-HSCT)
  * For subjects with DLBCL, PMBCL, and Gr3b-FL: relapsed or refractory disease following at least 2 prior regimens or following an auto-HSCT
  * For subjects with TH-FL: relapsed or refractory disease following at least 2 prior regimens or following an auto-HSCT. At least 1 prior regimen with an anti-CD20 mAb in combination with chemotherapy is required following documented transformation
  * For subjects with MCL (confirmed with cyclin D1 expression or evidence of t(11;14) by cytogenetics, fluorescent in situ hybridization (FISH) or PCR): relapsed or refractory disease after at least 1 prior regimen with chemo-immunotherapy (prior auto-HSCT is allowable)
* Karnofsky performance scale ≥ 60%
* Life expectancy of at least 6 months
* ANC > 1000/µL
* Platelet count > 50,000/µL
* For women of childbearing potential (defined as physiologically capable of becoming pregnant), agreement to use of highly effective contraception for at least 1 year following ACTR087 infusion. For men with partners of childbearing potential, agreement to use effective barrier contraception for at least 1 year following ACTR087 infusion

Exclusion Criteria:

* Known active central nervous system (CNS) involvement by malignancy. Subjects with prior CNS involvement with their lymphoma must have completed effective treatment of their CNS disease at least 3 months prior to enrollment with no evidence of disease clinically and at least stable findings on relevant CNS imaging
* Prior treatment as follows:

  * alemtuzumab within 6 months of enrollment
  * fludarabine, cladribine, or clofarabine within 3 months of enrollment
  * external beam radiation within 2 weeks of enrollment
  * mAb (including rituximab) within 2 weeks of enrollment
  * other lymphotoxic chemotherapy (including steroids except as below) within 2 weeks of enrollment
  * experimental agents within 3 half-lives prior to enrollment, unless progression is documented on therapy
* Serum creatinine ≥ 1.5 X age-adjusted upper limits of normal (ULN)
* Pulse oximetry < 92% on room air
* Direct bilirubin ≥ 3.0 mg/dL (50 mmol/L)
* Alanine transaminase (ALT) ≥ 3 times the ULN, unless determined to be directly due to lymphoma.
* Aspartate transaminase (AST) ≥ 3 times the ULN, unless determined to be directly due to lymphoma
* Class III or IV heart failure as defined by the New York Heart Association (NYHA), history of cardiac angioplasty or stenting, documented myocardial infarction or unstable angina within 6 months prior to enrollment, cardiac ejection fraction of < 45%, or other clinically significant cardiac disease
* Clinical history of, prior diagnosis of, or overt evidence of autoimmune disease, regardless of severity
* Clinically significant active infection, in the judgment of the investigator
* Pregnancy (negative serum pregnancy test to be obtained within 6 days prior to enrollment for subjects of childbearing potential)
* Breastfeeding
* Primary immunodeficiency
* Seropositive for Human Immunodeficiency Virus (HIV) 1 or HIV 2, or positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody
* Will need or has needed active treatment of a second malignancy within the prior 3 years before enrollment, other than FL, non-melanoma skin cancers, localized prostate cancer treated with curative intent, or cervical carcinoma in situ
* Is unable to receive any of the agents used in this study due a history of severe immediate hypersensitivity reaction (e.g. hypersensitivity to dimethyl sulfoxide (DMSO))
* History of prior allogeneic HSCT
* History of Richter's transformation from CLL
* Prior infusion of a genetically modified therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by dose limiting toxicities (DLTs) | 28 days
Safety as assessed by determination of the maximum tolerated dose (MTD) | 24 months
Safety as assessed by determination of the recommended phase 2 dose (RP2D) | 24 months
Safety as assessed by and adverse events, laboratory assessments and physical examinations | 24 months
Safety as assessed by mini-mental state examination (MMSE) | 24 months

SECONDARY OUTCOMES:
Overall response rate | 24 months
Duration of response | 24 months
Progression free survival | 24 months
Overall survival | 60 months

OTHER OUTCOMES:
ACRT087 persistence | 60 months
  Blood samples will be collected and analyzed for the presence of T-cells which express antibody coupled T-cell receptors, using flow cytometry and qPCR
Serum inflammatory markers | 169 days
Serum cytokine levels | 169 days
Rituximab serum concentrations | 147 days

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sachs, MD, Study Director — Cogent Biosciences, Inc.
Locations (7):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Yale University, New Haven, Connecticut
  - Loyola University Chicago, Maywood, Illinois
  - Indiana Bone and Marrow Transplantation, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338